CLINICAL TRIAL: NCT00985400
Title: Comparative Study of Oncologist Recommended, Home-Based Exercise Program and Relaxation Training for Physical Functioning and Symptom Control in Colon Cancer Patients
Brief Title: Doctor-Recommended Home-Based Exercise Program or Relaxation Training in Improving Physical Function and Controlling Symptoms in Patients With Stage IV or Recurrent Colon Cancer That Cannot Be Removed By Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2009-0288; MDA-2009-0288; CDR0000654446 (Other: NCI Clinical Trials); NCI-2011-02280 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2009-09-25; First posted 2009-09-28 (Estimated); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Colorectal Cancer
Keywords: recurrent colon cancer; stage IV colon cancer; Gastrointestinal; Exercise; Relaxation; Meditation
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Motor Activity | interventions — Resistance Training; Counseling; Surveys and Questionnaires; Relaxation Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise Program (Experimental): Arm I (exercise program): Oncologist advice; Resistance bands & pedometer with written/DVD instructions for resistance exercise twice a week for 16 weeks. Brief moderate-intensity walks multiple times a day for a total of 30 minutes increasing steps weekly by 10% to reach a minimum of 10,000 steps a day. Monthly newsletters; Telephone counseling weekly for 4 weeks then monthly for 12 weeks; and tailored message telephone prompts once every 2 weeks during last 12 weeks of the study intervention.
  Interventions: Behavioral: Exercise Program; Behavioral: Telephone-based intervention; Other: Counseling intervention; Other: Questionnaire administration
- Relaxation Intervention (Experimental): Arm II (relaxation program): Oncologist advice; Written/CD audio instructions on diaphragmatic breathing and guided imagery. Practice relaxation techniques for 15 minutes/day, 5-7 days/week, for 16 weeks. Monthly newsletters, telephone counseling, and tailored-message telephone prompts as in arm I.
  Interventions: Behavioral: Telephone-based intervention; Other: Counseling intervention; Other: Questionnaire administration; Behavioral: Relaxation Program

INTERVENTIONS:
Behavioral: Exercise Program — Resistance exercising using resistance bands 2 days per week, and brief moderate-intensity walks multiple times a day for a total of 30 minutes increasing steps weekly by 10% to reach a minimum of 10,000 steps a day
  Arms: Exercise Program
Behavioral: Telephone-based intervention — Patients will receive encouragement and social support from a telephone counselor once a week for the first 4 weeks and then once a month for the remaining 12 weeks.
Other: Counseling intervention — Patients will receive advice from their doctor (in person), physician assistant, or other midlevel provider about exercising. They will also be given this advice in a letter.
Other: Questionnaire administration
  Other Names: Survey
Behavioral: Relaxation Program — Relaxation techniques (breathing and meditation) provided at least 15 minutes per day for 5-7 days per week.
  Arms: Relaxation Intervention

SUMMARY:
The goal of this study is to compare the effects of exercise with the effects of relaxation training on physical function (how well participants perform normal daily activities) and symptoms related to your cancer diagnosis (such as tiredness, pain, and nausea).

DETAILED DESCRIPTION:
Study Groups:

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the flip of a coin) to 1 of 2 groups.

If you are in the exercise group, you will receive a doctor's recommendation to exercise (in-person advice and letters), newsletters on behavior change methods, resistance bands, a pedometer, and telephone counseling. A pedometer is a small device used to measure the number of steps you take.

If you are in the relaxation group, you will receive a doctor's recommendation to practice relaxation training (in-person advice and letters), newsletters on behavior change methods, written and video instructions for doing the relaxation techniques, and telephone counseling.

If you are in the Exercise Group:

* You will receive advice from your doctor (in person), physician's assistant, or other mid-level provider about exercising. You will be given advice on the use of your pedometer and resistance bands provided to you in this study, about the exercises provided and about keeping track of your progress on the exercise logs provided to you. You will also be given this advice in a letter.
* You will receive encouragement and support from a telephone counselor. The telephone counselor will contact you once a week for the first 4 weeks and then once a month for 12 weeks. The call will take about 5 minutes to complete.
* You will receive newsletters with stories about other cancer survivor experiences.
* You will be do resistance exercises using the resistance bands 2 days a week.

If you are in the Relaxation Group:

* You will receive advice from your doctor (in person), physician's assistant or other mid-level provider about relaxation techniques. You will be given advice on practicing the breathing and meditation techniques provided to you in this study, on how long and how often you are performing your relaxation techniques, and on keeping track of your relaxation practice on the relaxation logs provided to you. -You will also be given this advice in a letter.
* You will receive encouragement and support from a telephone counselor. The telephone counselor will contact you once a week for the first 4 weeks and then once a month for 12 weeks. The call will take about 5 minutes to complete.
* You will receive newsletters with stories about other cancer survivor experiences.
* You will be perform the relaxation techniques at least 15 minutes a day for 5-7 days a week.

All participants will continue the group exercises or relaxation techniques for 16 weeks.

Follow-Up Visit:

You will have a follow-up visit during Weeks 16-20. At this visit, you will complete the following tests and procedures:

* Your medical history will be recorded.
* Your performance status will be recorded.
* You will complete the 11 questionnaires.
* You will complete the exercise tests to measure how your body uses oxygen, to test your lower body strength, to test your upper body strength, and to test your flexibility and balance.

Length of Study:

You will remain on study for 16-20 weeks.

This is an investigational study.

Up to 154 patients will take part in this multicenter study. Up to 154 may be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of stage IV or recurrent colorectal cancer
2. Age >/= 18 years
3. ECOG performance status of 0 -1
4. Able to communicate in English or Spanish
5. Able to give informed consent
6. Adequate organ function -Total bilirubin < 1.5 x the institutional upper-normal limits (IUNL); AST (SGOT) and/or ALT (SGPT) < 2.5 x IUNL; Patients with liver metastasis AST/ (SGOT) and/or ALT (SGPT) < 5 x IUNL
7. Adequate bone marrow function: - Absolute neutrophil count > 1,000/microLiters; Platelets > 50,000/microLiters
8. Able to ambulate without assistance
9. Has access to a telephone in order to receive pre-recorded telephone messages and for multiple counseling sessions.

Exclusion Criteria:

1. Major surgery in the past 8 weeks
2. Medical contraindications to home-based exercise as defined by the treating physician
3. Symptomatic Bone Metastases
4. Unstable Angina (current symptomatic angina at time of enrollment)
5. Class III/IV heart failure according to NYHA classification system
6. Pulmonary conditions that require oxygen
7. Unable to ambulate without assistance (cane, walker, etc)
8. Exercising at a moderate-vigorous intensity for 150 minutes or more per week, exercising at a vigorous intensity for more than 20 minutes on 3 or more days per week, or performing resistance exercises for more than 20 minutes per day on two or more days per week for 3 months or more.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2010-11-05 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | 3 year study period
Patient retention | 3 year study period
Program and assessment implementation | 3 year study period
Patient adherence to behavioral recommendations | Up to 20 weeks
Effect size of the exercise intervention on physical function | Up to 20 weeks

SECONDARY OUTCOMES:
Effect size of the exercise intervention on symptoms and quality of life | Up to 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Karen Basen-Engquist, PhD, Study Chair — M.D. Anderson Cancer Center; Michael J. Fisch, MD, MPH, FACP, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — https://clinicaltrials.gov/ct2/show/NCT00985400?term=2009-0288&draw=2&rank=1
- See also: University of Texas MD Anderson Cancer Center Official Website — http://www.mdanderson.org